CLINICAL TRIAL: NCT00998075
Title: A Phase I, Open-Label, Randomized, Single-Centre, 3-Way Crossover Bioequivalence Study Comparing a Fixed Dose Combination Capsule of Esomeprazole 40 mg and Acetylsalicylic Acid 325 mg With Free Combinations of Esomeprazole Capsule 40 mg and Acetylsalicylic Acid Tablet 325 mg and Esomeprazole Tablet
Brief Title: Study Comparing Esomeprazole and Acetylsalicylic Acid (ASA) Combined Together as One Capsule Versus These Medications Taken Separately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D961FC00007
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Peptic Ulcer Disease
Keywords: Bioequivalence; ASA; Esomeprazole; peptic ulcer disease; primary cardiovascular protection; healthy volunteers
MeSH Terms: conditions — Peptic Ulcer | interventions — Esomeprazole; Aspirin

ARMS (3):
- 1 (Active Comparator): Esomeprazole 40 mg/ASA 325 mg Fixed Dose Combination Capsule
  Interventions: Drug: Esomeprazole/ASA Fixed Combination
- 2 (Active Comparator): Esomeprazole Clinical Trial Capsule 40 mg and 1 Aspirin® Non Enteric Coated Immediate Release Tablet 325 mg
  Interventions: Drug: Esomeprazole - Nexium; Drug: ASA
- 3 (Active Comparator): Esomeprazole MUPS Tablet 40 mg and 1 Aspirin® Non Enteric Coated Immediate Release Tablet 325 mg
  Interventions: Drug: Esomeprazole - Nexium; Drug: ASA

INTERVENTIONS:
Drug: Esomeprazole/ASA Fixed Combination — Capsule, oral, single dose
  Arms: 1
Drug: Esomeprazole - Nexium — Clinical Trial Capsule or MUPS Tablet, oral, single dose
  Arms: 2; 3
Drug: ASA — Tablet, oral, single dose
  Other Names: Aspirin
  Arms: 2; 3

SUMMARY:
The purpose of this study is to investigate whether treatment with a combination capsule of Esomeprazole 40 mg and Aspirin (ASA) 325 mg is bioequivalent (i.e.has the same effect within the body) as these medications taken separately. Two different forms of esomeprazole (tablets and capsules) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female within the age range of 20 to 50 years
* Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 29.9 kg/m2

Exclusion Criteria:

* Documented upper gastrointestinal surgery
* Use of any proton pump inhibitors or any bismuth preparations (e.g. Pepto-Bismol®) within 14 days preceding the screening visit

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration-time curve from time 0 to the last quantifiable concentration for esomeprazole administered as fixed dose combination (FDC) to esomeprazole administered as free combinations | PK samples to be taken for bioanalysis over a 24-hour period following dosing on Day 1 of Period I and Day 1 of Period II and III.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Total area under the plasma concentration-time curve (AUC0-inf), AUC0-t, Cmax, time to Cmax (Tmax), and half-life (t½) of esomeprazole | PK samples to be taken for bioanalysis over a 24-hour period following dosing for each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: TJørgen Næsdal, MD, PhD, Study Director — AstraZeneca R&D; Pierre Geoffroy, M.D. C.M., M.S, Principal Investigator — Biovail Contract Research (BCR)a Division of Biovail Corporation
Locations (1):
- Research Site, Scarborough Village, Ontario, Canada